CLINICAL TRIAL: NCT04815200
Title: Efficiency of Using Copper-Nickel-Titanium Versus Nickel-Titanium Arch Wires on Anterior Segment Crowding Alleviation in Group of Adults With Moderate Crowding: A Randomized Controlled Clinical Trial
Brief Title: Efficiency of Using Copper-Nickel-Titanium Versus Nickel-Titanium Arch Wires on Anterior Segment Crowding Alleviation in Group of Adults With Moderate Crowding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Bedir Abd El Hady El Gendy, master student, department of orthodontics, Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25121
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Crowding of Anterior Mandibular Teeth

STUDY DESIGN:
Intervention Model Description: Patient will receive 0.014 round Copper Nickel titanium CuNiTi archwire and will be ligated using a ligature wire
Masking Description: i) To participant (subjects): Patients can be blinded as they do not know the type of wire used. ii) To Assessor: The assessor (different than the main operator) will carry out the measurements blindly on the pre and post models.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nickel titanium NiTi arch wire (Gold Standard, control group) (Other): Patient will receive 0.014 round Nickel titanium NiTi archwire and will be ligated using a ligature wire with Follow up for 2 months.
  Interventions: Device: Copper Nickel titanium arch wire

INTERVENTIONS:
Device: Copper Nickel titanium arch wire — Patient will receive 0.014 round Copper Nickel titanium CuNiTi archwire and will be ligated using a ligature wire.
  Other Names: CuNiTi

SUMMARY:
Evaluate the efficiency of using copper nickel titanium (CuNiTi) arch wire on the initial stage of leveling and alignment regarding their rate of alignment in comparison to Conventional Nickel Titanium arch wire (NiTi) by Measuring the amount and rate of alignment achieved every 2 weeks for a period of 2 months.

.

DETAILED DESCRIPTION:
Leveling and alignment is the first stage in fixed orthodontic treatment, performed for every patient. Copper nickel titanium (CuNiTi) was modified from conventional nickel titanium (NiTi) to stabilize the super elasticity properties of the initial nickel titanium (NiTi) arch wire against cyclic deformation. The addition of copper to traditional nickel titanium enhances thermal reactive properties and consistency of forces.so the aim of the study is to Evaluate the efficiency of using copper nickel titanium (CuNiTi) arch wire on the initial stage of leveling and alignment regarding their rate of alignment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged (18~33).
2. Moderate crowding (4-8)10.
3. No extractions required.

Exclusion Criteria:

1. Previous orthodontic treatment.
2. Missing teeth other than the wisdoms.
3. Patient with dental anomalies.
4. Patient having a deep bite, open bite or cross bite.

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-18 (Estimated); Primary Completion 2022-03-18 (Estimated); Study Completion 2022-04-18 (Estimated)

PRIMARY OUTCOMES:
Rate of alignment. | 8 weeks
  Measuring the amount and rate of alignment of teeth which achieved every 2 weeks for a period of 8 weeks using (mm) as numerical unit of measurement and method of measurement is '' Little's irregularity index''

SECONDARY OUTCOMES:
inter-canine arch perimeter width | 8 weeks
  measure inter canine perimeter width every 2 weeks using Unit of measurement numerical (mm) though ortho analyzer 3shape software
pain assessed by NRS | first 24 hours
  measuring pain associated after placement of the wire through printed copy of numerical rating pain scale with a person rates their pain on a scale of 0 to 10,Zero means "no pain," while 10 means "the worst possible pain."
inter-molar arch perimeter width. | 8 weeks
  measure inter-molar arch perimeter width every 2 weeks using a numerical unit of measurement (mm) through ortho analyzer 3shape software

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided